CLINICAL TRIAL: NCT03048851
Title: Immediate and Maintaining Efficacy of New Protocols in the Treatment of Upper Limb Dysfunctions in Patients With Cerebral Palsy
Brief Title: Efficacy of New Protocols in the Treatment of Upper Limb Dysfunctions in Patients With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 103-7425A3
Record Dates: First submitted 2016-10-10; First posted 2017-02-09 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2019-08

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; sensory electrical stimulation; virtual reality constraint-induced therapy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Low dosage SES group (Experimental): Low dosage SES group received the low dosage SES training in addition to traditional rehabilitation. Each SES session involved electrical stimulation followed by UE training in addition to home program.
  Interventions: Device: Low dosage SES group
- High dosage SES group (Experimental): High dosage SES group received the high dosage SES training in addition to traditional rehabilitation. Each SES session involved electrical stimulation followed by UE training in addition to home program.
  Interventions: Device: High dosage SES group
- VRCIT group (Experimental): VRCIT group received the VRCIT training in addition to traditional rehabilitation.Each VRCIT session involved practice of functional tasks with the more affected UE followed by virtual-reality based eye-hand coordination tasks with the more affected UE for, in addition to home program, and restraint of the less affected UE for 1.5 hours per day.
  Interventions: Device: VRCIT group
- VRCIT+SES group (Experimental): VRCIT+SES group received the VRCIT and SES training in addition to traditional rehabilitation.
  Interventions: Device: VRCIT+SES group
- traditional rehabilitation group (Active Comparator): Shame control group received the shame SES and traditional rehabilitation programs.
  Interventions: Procedure: traditional rehabilitation program

INTERVENTIONS:
Device: Low dosage SES group — The participants were randomly assigned to one of the five intervention groups. Low dosage SES group received the SES (Micro-Z Mini, Prizm Medical Inc., USA) training in addition to traditional rehabilitation. Each SES session involved electrical stimulation followed by UE training in addition to home program.The novel SES programs were conducted twice per week, for 12 weeks. Each SES session involved electrical stimulation followed by UE training in addition to home program. The SES was applied to the forearm and whole hand with mesh glove (Electro-Mesh Glove-Sleeve Electrode Kit) for 45 minutes and arm with wrap for 45 minutes. The pulse width was set to 300us for all stimulation levels. The frequency was set to 100 Hz and 10 Hz.
  Other Names: novel sensory electrical stimulation program
  Arms: Low dosage SES group
Device: High dosage SES group — The participants were randomly assigned to one of the five intervention groups. High dosage SES group received the SES (Micro-Z Mini, Prizm Medical Inc., USA) training in addition to traditional rehabilitation. Each SES session involved electrical stimulation followed by UE training in addition to home program.The novel SES programs were conducted twice per week, for 12 weeks. Each SES session involved electrical stimulation followed by UE training in addition to home program. The SES was applied to the forearm and whole hand with mesh glove (Electro-Mesh Glove-Sleeve Electrode Kit) for 90 minutes and arm with wrap for 90 minutes. The pulse width was set to 300us for all stimulation levels. The frequency was set to 100 Hz and 10 Hz.
  Other Names: novel sensory electrical stimulation program
  Arms: High dosage SES group
Device: VRCIT group — The participants were randomly assigned to one of the five intervention groups. VRCIT group received the VRCIT training plus traditional rehabilitation, conducted twice per week for 12 weeks. Each VRCIT session involved practice of functional tasks with the more affected UE followed by virtual-reality based eye-hand coordination tasks with the more affected UE for, plus home program, and restraint of the less affected UE for 1.5 hours per day. The functional training of the more affected UE focused on massive practice of functional activities using the more affected arm, with the principles of shaping and repetitive task practice applied during training. The VRCIT combined CIT and commercially available VR-based systems including Sony Playstation EyeToy and Nintendo Wii.
  Other Names: virtual reality based Constraint-induced therapy
  Arms: VRCIT group
Device: VRCIT+SES group — The participants were randomly assigned to one of the five intervention groups. VRCIT+SES group executed VR programs by affected UE in Mesh-gloves (Electro-Mesh Glove-Sleeve Electrode Kit) with the optimal SES (Micro-Z Mini, Prizm Medical Inc., USA) protocol formulated from the 1st phase study. The VRCIT program was conducted 1.5 hours/time, twice/week for 12 weeks. The VRCIT combined CIT and commercially available VR-based systems. Some commercially programs, such as Sony Playstation EyeToy (Sony Computer Entertainment America, Foster City, Calif., USA), and Nintendo Wii (Nintendo Domestic Distributor, College Point, N.Y., USA).
  Other Names: combined VR based Constraint-induced therapy & SES
  Arms: VRCIT+SES group
Procedure: traditional rehabilitation program — The participants were randomly assigned to one of the five intervention groups. The absence of muscle contractions was controlled by the investigator the sham stimulation was carried out identically, but the stimulation amplitude was set to 0 milliampere(mA). Subjects were not informed about the stimulation level and were instructed to distract attention from the stimulation.
  Arms: traditional rehabilitation group

SUMMARY:
Immediate and maintaining Efficacy of new protocols in the treatment of upper limb dysfunctions in patients with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common childhood motor disability. Spasticity and loss of dexterity are the major problems for motor disability of upper extremity (UE) in patients with CP. This study propose two novel treatment protocols: sensory electrical stimulation (SES) and virtual reality constraint-induced therapy (VRCIT) to improve function of UE in patients with CP. Investigators hypothesize that combined SES and VRCIT treatment have better effect than single therapy (SES or VRCIT).

ELIGIBILITY:
* Inclusion Criteria:

  * Diagnosis with spastic CP with Gross Motor Function Classification System(GMFCS) levels I-IV
  * Aged 2-24 years
  * Ability to undergo clinical assessment
  * Ability to comprehend commands and cooperate during an examination
* Exclusion Criteria:

  * Chromosomal abnormalities
  * Progressive neurological disorder or severe concurrent illness or disease not typically associated with CP
  * Active medical conditions such as pneumonia or poor physical conditions that would interfere with participation
  * Any major surgery or nerve block in the preceding 3 months
  * Metabolic or hormonal disturbance
  * Cardiovascular disorder
  * Poor tolerance or a poor cooperation during assessment

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2015-08; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
change from baseline of muscle tone and basic motor abilities of the upper limb muscles in 12 and 24 weeks | baseline, 12weeks, 24weeks
  Muscle tone of the upper limb muscles assessment by Modified Ashworth Scale and Myoton (© 2011 Myoton AS.). Basic motor abilities included the assessments of the Bruininks-Oseretsky Test of Motor Proficiency II (BOT II), Melbourne Assessment 2 (MA2), Quality of upper extremity skills test (QUEST). The measure is a composite.

SECONDARY OUTCOMES:
change from baseline of quality of life in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The health-related quality of life(HRQOL) assess by Cerebral Palsy Quality of Life (CP QOL) for Child and adolescent. The CP QOL is a measure of HRQOL specific to children and adolescent with cerebral palsy.
change from baseline of activities of daily living (ADL) in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The ADL assessments included Functional Independence Measure for Children (WeeFIM) and Pediatric Motor Activity Log (PMAL). The measure is a composite.
change from baseline of bone mineral density in 12 and 24 weeks | baseline, 12weeks, 24weeks
  he areal bone mineral density (aBMD) (g/cm2) will be measured at the lumbar spine (L1 to L4) and the humerus of the more-affected limb using dual X-ray absorptiometry (DXA).
change from baseline of Metabolism and Body composition in 12 and 24 weeks | baseline, 12weeks, 24weeks
  The measure included the total energy expenditure (kcal/min), active energy expenditure (kcal/min), total number of steps, physical activity levels and duration, sleep duration and efficiency, weight, total body water, skeletal muscle mass (SMM), body fat mass (BFM), fat free mass, percent body fat, waist-hip ratio (WHR), and basal metabolic rate (BMR) by the devices of SenseWear(© 2013 BodyMedia, Inc.) and Body Composition Analyzer(InBody230). The measure is a composite.
change from baseline of kinematic analysis in 12 and 24 weeks | baseline, 12weeks, 24weeks
  Kinematic analysis for patients performing Reach-to-grasp and Eye-hand coordination tasks.The measure is a composite.
change from baseline of muscle strength and endurance in 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  The device (Hoggan-5081) for kinetic analysis combined range of motion (ROM), muscle testing (MicroFET3) and grip and pinch gauge (MicroFET4) and data capture software, attached to a computer for more thorough testing. MicroFET4 combined pinch gauge and grip tester in a single device with high test-retest reliability. The Grip Test included Maximum Grip Test, 5 Position Grip Test, Rapid Exchange Grip Test, Hand Grip Fatigue Test. The Pinch Test included key Pinch, palmar Pinch, and tip pinch. MicroFET3 combined Muscle Tester and ROM Gauge. Peak force and average strength were obtained. The padded attachment that was fit in the palm of the hand allowed the administrators to provide direct resistance to movement of the extremity. For arm strength test, the examiner manually stabilized the body parts proximal to the tested limb segment during testing and asked participants to exert a maximal isometric muscle contraction lasting 3-seconds while the dynamometer was held stationary.
change from baseline of severity in 12 and 24 weeks | baseline, 12 weeks, 24 weeks
  The severity is evaluated by Gross Motor Function Classification System(GMFCS), Manual Ability Classification System (MACS).The assessments for body function included Modified Ashworth Scale (MAS), strength, endurance, and trunk and limb involvement, etc. The measure is a composite.
change from baseline of reaction-time in 12 and 24 weeks | baseline, 12 weeks ,24 weeks
  To examine the reaction time by CANTAB® software.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD,PhD, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No